CLINICAL TRIAL: NCT00080171
Title: Osteoarthritis Initiative (OAI): A Knee Health Study
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: GlaxoSmithKline (Industry); Merck Sharp & Dohme LLC (Industry); Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NIAMS-109
Record Dates: First submitted 2004-03-24; First posted 2004-03-25 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2009-03

CONDITIONS: Osteoarthritis; Knee Osteoarthritis
Keywords: Osteoarthritis; Knee Pain; Knee Health
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine

SUMMARY:
Knee osteoarthritis (OA) is the most common cause of disability in adults. The "Osteoarthritis Initiative (OAI): A Knee Health Study" is a nationwide research study that will help researchers gather more information about the physical changes that occur prior to the onset of arthritis symptoms or before OA gets worse. The purpose of this study is to examine people who have knee OA or are at high risk for knee OA; information will be used to better understand how to prevent and treat knee OA.

DETAILED DESCRIPTION:
Knee OA causes more health problems and medical expenses that any other form of arthritis. Symptoms of OA can range from stiffness and mild pain to severe joint pain and even disability. Previous research has shown that certain factors, such as knee pain, prior knee injury or knee surgery, OA of the hand, or obesity, may lead to knee OA. The OAI is a multicenter, observational study of knee OA that will collect information on potential biomarkers for OA and trends in OA onset and progression.

The OAI will recruit and follow participants who have knee OA or are at high risk for developing knee OA for an eight-year period at one of four clinical centers. Blood and urine collection, magnetic resonance imaging (MRI), and X-rays will be completed at each of four annual follow-up visits. A questionnaire and physical examination at screening will assess for risk factors for the development and progression of knee OA. Levels of knee pain and physical disability will be assessed at study start and at each of the follow-up visits by questionnaire and examination.

ELIGIBILITY:
Inclusion Criteria:

Must meet one of the following criteria:

* Overweight
* Previous knee injury or surgery
* Knee pain during the past year. Participants do not need to have current knee pain to take part in the study.
* Parent or sibling who had knee replacement

Exclusion Criteria:

* Rheumatoid arthritis
* Joint replacements in both knees
* Unable to walk without assistance
* Unable to undergo MRI of the knee

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have knee OA or are at high risk for developing knee OA
Sampling Method: Non-Probability Sample
Enrollment: 4796 (Actual)
Dates: Start 2004-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Lester, PhD, Study Director — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (5):
- United States (5):
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island / Brown University, Pawtucket, Rhode Island

REFERENCES:
- [Derived] Eckstein F, Chaudhari AS, Hunter DJ, Wirth W. Comparison between coronal FLASH and sagittal double echo steady state MRI in detecting longitudinal cartilage thickness change by fully automated segmentation - Data from the FNIH biomarker cohort. Osteoarthr Cartil Open. 2025 Aug 5;7(3):100657. doi: 10.1016/j.ocarto.2025.100657. eCollection 2025 Sep. PMID 40822965
- [Derived] Tore NG, Liles S, Werner DM, Cleveland RJ, Bye TV, Golightly Y, Jakiela JT, White DK. The relation of activity patterns with incident slow gait speed over 4 years in adults with knee osteoarthritis: Data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2025 Sep;33(9):1121-1129. doi: 10.1016/j.joca.2025.06.002. Epub 2025 Jun 6. PMID 40484272
- [Derived] Bharadwaj UU, Lynch JA, Joseph GB, Akkaya Z, Nevitt MC, Lane NE, McCulloch CE, Link TM. Intra-articular Knee Injections and Progression of Knee Osteoarthritis: Data from the Osteoarthritis Initiative. Radiology. 2025 May;315(2):e233081. doi: 10.1148/radiol.233081. PMID 40423542
- [Derived] Moradi K, Mohammadi S, Roemer FW, Momtazmanesh S, Hathaway Q, Ibad HA, Hunter DJ, Guermazi A, Demehri S. Progression of Bone Marrow Lesions and the Development of Knee Osteoarthritis: Osteoarthritis Initiative Data. Radiology. 2024 Sep;312(3):e240470. doi: 10.1148/radiol.240470. PMID 39287521
- [Derived] Wirth W, Maschek S, Wisser A, Eder J, Baumgartner CF, Chaudhari A, Berenbaum F, Eckstein F; OA-BIO Consortium. Evaluation of an automated laminar cartilage T2 relaxation time analysis method in an early osteoarthritis model. Skeletal Radiol. 2025 Mar;54(3):571-584. doi: 10.1007/s00256-024-04786-1. Epub 2024 Sep 4. PMID 39230576
- [Derived] Zhang H, Shuai T, Wang J, Li K, Nie Y. Relationship Between 2 Years of Muscle Strength Decrease and Volume Loss of Menisci and Cartilage According to Knee Pain in Mild and Moderate Knee Osteoarthritis. Am J Phys Med Rehabil. 2024 Jan 1;104(1):1-7. doi: 10.1097/PHM.0000000000002507. Epub 2024 Apr 30. PMID 38686814
- [Derived] Li M, Nie Y, Zeng Y, Wu Y, Wu L, Liu Y, Shen B. Eight-year trajectories of malalignment progression in symptomatic knee osteoarthritis. Chin Med J (Engl). 2022 Nov 5;135(21):2570-2576. doi: 10.1097/CM9.0000000000002044. PMID 36583920
- [Derived] Wirth W, Maschek S, Wisser A, Guermazi A, Hunter DJ, Kwoh CK, Nevitt MC, Eckstein F, Roemer FW. Selection of Knees With Subsequent Cartilage Thickness Loss Based on Magnetic Resonance Imaging Semiquantitative Grading: Data From the Osteoarthritis Initiative Foundation for the National Institutes of Health Biomarker Cohort. Arthritis Care Res (Hoboken). 2023 Aug;75(8):1773-1782. doi: 10.1002/acr.25078. Epub 2023 Feb 22. PMID 36576026
- [Derived] Mohajer B, Dolatshahi M, Moradi K, Najafzadeh N, Eng J, Zikria B, Wan M, Cao X, Roemer FW, Guermazi A, Demehri S. Role of Thigh Muscle Changes in Knee Osteoarthritis Outcomes: Osteoarthritis Initiative Data. Radiology. 2022 Oct;305(1):169-178. doi: 10.1148/radiol.212771. Epub 2022 Jun 21. PMID 35727152
- [Derived] Li J, Fu S, Gong Z, Zhu Z, Zeng D, Cao P, Lin T, Chen T, Wang X, Lartey R, Kwoh CK, Guermazi A, Roemer FW, Hunter DJ, Ma J, Ding C. MRI-based Texture Analysis of Infrapatellar Fat Pad to Predict Knee Osteoarthritis Incidence. Radiology. 2022 Sep;304(3):611-621. doi: 10.1148/radiol.212009. Epub 2022 May 31. PMID 35638929
- [Derived] Lee JJ, Namiri NK, Astuto B, Link TM, Majumdar S, Pedoia V. Personalized Risk Model and Leveraging of Magnetic Resonance Imaging-Based Structural Phenotypes and Clinical Factors to Predict Incidence of Radiographic Osteoarthritis. Arthritis Care Res (Hoboken). 2023 Mar;75(3):501-508. doi: 10.1002/acr.24877. Epub 2022 Dec 10. PMID 35245407
- [Derived] Steidle-Kloc E, Dannhauer T, Wirth W, Eckstein F. Responsiveness of Subcutaneous Fat, Intermuscular Fat, and Muscle Anatomical Cross-Sectional Area of the Thigh to Longitudinal Body Weight Loss and Gain: Data from the Osteoarthritis Initiative (OAI). Cells Tissues Organs. 2022;211(5):555-564. doi: 10.1159/000520037. Epub 2021 Oct 7. PMID 34619678
- [Derived] Canton G, Hippe DS, Chen L, Waterton JC, Liu W, Watase H, Balu N, Sun J, Hatsukami TS, Yuan C. Atherosclerotic Burden and Remodeling Patterns of the Popliteal Artery as Detected in the Magnetic Resonance Imaging Osteoarthritis Initiative Data Set. J Am Heart Assoc. 2021 Jun;10(11):e018408. doi: 10.1161/JAHA.120.018408. Epub 2021 May 17. PMID 33998279
- [Derived] Fuerst D, Wirth W, Gaisberger M, Hunter DJ, Eckstein F. Association of Superficial Cartilage Transverse Relaxation Time With Osteoarthritis Disease Progression: Data From the Foundation for the National Institutes of Health Biomarker Study of the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2022 Nov;74(11):1888-1893. doi: 10.1002/acr.24627. Epub 2022 Jul 12. PMID 33973402
- [Derived] Hu B, Han D, Nevitt MC, Wise BL, Segal NA. Longitudinal Relationship Between Physical Activity and Joint Space Narrowing: Forty-Eight-Month Follow-Up Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2022 Jul;74(7):1163-1171. doi: 10.1002/acr.24554. Epub 2022 Apr 13. PMID 33411980
- [Derived] Eckstein F, Chaudhari AS, Fuerst D, Gaisberger M, Kemnitz J, Baumgartner CF, Konukoglu E, Hunter DJ, Wirth W. Detection of Differences in Longitudinal Cartilage Thickness Loss Using a Deep-Learning Automated Segmentation Algorithm: Data From the Foundation for the National Institutes of Health Biomarkers Study of the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2022 Jun;74(6):929-936. doi: 10.1002/acr.24539. Epub 2022 Apr 1. PMID 33337584
- [Derived] Campbell TM, Ramsay T, Trudel G. Knee Flexion Contractures Are Associated with Worse Pain, Stiffness, and Function in Patients with Knee Osteoarthritis: Data from the Osteoarthritis Initiative. PM R. 2021 Sep;13(9):954-961. doi: 10.1002/pmrj.12497. Epub 2020 Nov 10. PMID 32969154
- [Derived] Roth M, Emmanuel K, Wirth W, Kwoh CK, Hunter DJ, Hannon MJ, Eckstein F. Changes in Medial Meniscal Three-Dimensional Position and Morphology As Predictors of Knee Replacement in Rapidly Progressing Knee Osteoarthritis: Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2021 Jul;73(7):1031-1037. doi: 10.1002/acr.24193. PMID 32198847
- [Derived] Haj-Mirzaian A, Mohajer B, Guermazi A, Conaghan PG, Lima JAC, Blaha MJ, Bingham CO, Roemer FW, Cao X, Demehri S. Statin Use and Knee Osteoarthritis Outcome Measures according to the Presence of Heberden Nodes: Results from the Osteoarthritis Initiative. Radiology. 2019 Nov;293(2):396-404. doi: 10.1148/radiol.2019190557. Epub 2019 Sep 10. PMID 31502936
- [Derived] Ruhdorfer A, Wirth W, Culvenor AG, Eckstein F. Reduction in Thigh Muscle Strength Occurs Concurrently but Does Not Seem to Precede Incident Knee Pain in Women: Data From the Osteoarthritis Initiative Cohort. Am J Phys Med Rehabil. 2020 Jan;99(1):33-40. doi: 10.1097/PHM.0000000000001271. PMID 31343500
- [Derived] Wirth W, Maschek S, Roemer FW, Sharma L, Duda GN, Eckstein F. Radiographically normal knees with contralateral joint space narrowing display greater change in cartilage transverse relaxation time than those with normal contralateral knees: a model of early OA? - data from the Osteoarthritis Initiative (OAI). Osteoarthritis Cartilage. 2019 Nov;27(11):1663-1668. doi: 10.1016/j.joca.2019.06.013. Epub 2019 Jul 10. PMID 31301430
- [Derived] Eckstein F, Maschek S, Roemer FW, Duda GN, Sharma L, Wirth W. Cartilage loss in radiographically normal knees depends on radiographic status of the contralateral knee - data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2019 Feb;27(2):273-277. doi: 10.1016/j.joca.2018.10.006. Epub 2018 Oct 28. PMID 30394330
- [Derived] Bricca A, Wirth W, Juhl CB, Kemnitz J, Hunter DJ, Kwoh CK, Eckstein F, Culvenor AG. Moderate Physical Activity and Prevention of Cartilage Loss in People With Knee Osteoarthritis: Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2019 Feb;71(2):218-226. doi: 10.1002/acr.23791. PMID 30339323
- [Derived] Jacobs CA, Vranceanu AM, Thompson KL, Lattermann C. Rapid Progression of Knee Pain and Osteoarthritis Biomarkers Greatest for Patients with Combined Obesity and Depression: Data from the Osteoarthritis Initiative. Cartilage. 2020 Jan;11(1):38-46. doi: 10.1177/1947603518777577. Epub 2018 Jun 1. PMID 29855190
- [Derived] Hu B, Skou ST, Wise BL, Williams GN, Nevitt MC, Segal NA. Lower Quadriceps Rate of Force Development Is Associated With Worsening Physical Function in Adults With or at Risk for Knee Osteoarthritis: 36-Month Follow-Up Data From the Osteoarthritis Initiative. Arch Phys Med Rehabil. 2018 Jul;99(7):1352-1359. doi: 10.1016/j.apmr.2017.12.027. Epub 2018 Jan 31. PMID 29408538
- [Derived] Wirth W, Hunter DJ, Nevitt MC, Sharma L, Kwoh CK, Ladel C, Eckstein F. Predictive and concurrent validity of cartilage thickness change as a marker of knee osteoarthritis progression: data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2017 Dec;25(12):2063-2071. doi: 10.1016/j.joca.2017.08.005. Epub 2017 Aug 31. PMID 28838858
- [Derived] Steidle-Kloc E, Culvenor AG, Dorrenberg J, Wirth W, Ruhdorfer A, Eckstein F. Relationship Between Knee Pain and Infrapatellar Fat Pad Morphology: A Within- and Between-Person Analysis From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2018 Apr;70(4):550-557. doi: 10.1002/acr.23326. Epub 2018 Mar 11. PMID 28704603
- [Derived] Kemnitz J, Wirth W, Eckstein F, Ruhdorfer A, Culvenor AG. Longitudinal change in thigh muscle strength prior to and concurrent with symptomatic and radiographic knee osteoarthritis progression: data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2017 Oct;25(10):1633-1640. doi: 10.1016/j.joca.2017.07.003. Epub 2017 Jul 8. PMID 28698106
- [Derived] Veronese N, Stubbs B, Noale M, Solmi M, Vaona A, Demurtas J, Nicetto D, Crepaldi G, Schofield P, Koyanagi A, Maggi S, Fontana L. Fried potato consumption is associated with elevated mortality: an 8-y longitudinal cohort study. Am J Clin Nutr. 2017 Jul;106(1):162-167. doi: 10.3945/ajcn.117.154872. Epub 2017 Jun 7. PMID 28592612
- [Derived] Wirth W, Maschek S, Beringer P, Eckstein F. Subregional laminar cartilage MR spin-spin relaxation times (T2) in osteoarthritic knees with and without medial femorotibial cartilage loss - data from the Osteoarthritis Initiative (OAI). Osteoarthritis Cartilage. 2017 Aug;25(8):1313-1323. doi: 10.1016/j.joca.2017.03.013. Epub 2017 Mar 27. PMID 28351705
- [Derived] Veronese N, Stubbs B, Noale M, Solmi M, Luchini C, Maggi S. Adherence to the Mediterranean diet is associated with better quality of life: data from the Osteoarthritis Initiative. Am J Clin Nutr. 2016 Nov;104(5):1403-1409. doi: 10.3945/ajcn.116.136390. Epub 2016 Sep 28. PMID 27680996
- [Derived] Collins JE, Deshpande BR, Katz JN, Losina E. Race- and Sex-Specific Incidence Rates and Predictors of Total Knee Arthroplasty: Seven-Year Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2016 Jul;68(7):965-73. doi: 10.1002/acr.22771. PMID 26554629
- [Derived] Eckstein F, Collins JE, Nevitt MC, Lynch JA, Kraus VB, Katz JN, Losina E, Wirth W, Guermazi A, Roemer FW, Hunter DJ; FNIH OA Biomarkers Consortium. Brief Report: Cartilage Thickness Change as an Imaging Biomarker of Knee Osteoarthritis Progression: Data From the Foundation for the National Institutes of Health Osteoarthritis Biomarkers Consortium. Arthritis Rheumatol. 2015 Dec;67(12):3184-9. doi: 10.1002/art.39324. PMID 26316262
- [Derived] Eckstein F, Kwoh CK, Link TM; OAI investigators. Imaging research results from the osteoarthritis initiative (OAI): a review and lessons learned 10 years after start of enrolment. Ann Rheum Dis. 2014 Jul;73(7):1289-300. doi: 10.1136/annrheumdis-2014-205310. Epub 2014 Apr 12. PMID 24728332
- [Derived] Baum T, Joseph GB, Arulanandan A, Nardo L, Virayavanich W, Carballido-Gamio J, Nevitt MC, Lynch J, McCulloch CE, Link TM. Association of magnetic resonance imaging-based knee cartilage T2 measurements and focal knee lesions with knee pain: data from the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2012 Feb;64(2):248-55. doi: 10.1002/acr.20672. PMID 22012846
- See also: Click here for the Osteoarthritis Initiative [OAI] Web site. — http://www.oai.ucsf.edu